CLINICAL TRIAL: NCT00816777
Title: Feasibility and Prospective Randomized Study of Transarterial Chemoembolization Using Irinotecan Bead in Combination With Second Line Chemotherapy in the Treatment of Patients With Unresectable Metastatic Colorectal Cancer
Brief Title: Chemoembolization, Irinotecan Bead, Second Line Chemotherapy Treatment of Unresectable Metastatic Colorectal Cancer
Acronym: PARAGON
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Generic Devices Consulting, Inc. (Industry)
Collaborators: Biocompatibles UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA1013; IDE G070122 (Other: FDA IDE)
Record Dates: First submitted 2009-01-02; First posted 2009-01-05 (Estimated); Results first posted 2015-09-18 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-02

CONDITIONS: Unresectable Metastatic Colo-rectal Cancer
Keywords: Cancer; Carcinoma; Colon Cancer; Colorectal Cancer; Gastric Cancer; Gastrointestinal Cancer; Metastases; Metastatic Cancer; Metastatic Colorectal Cancer; Oncology; Rectal Cancer
MeSH Terms: conditions — Neoplasms; Carcinoma; Colonic Neoplasms; Colorectal Neoplasms; Stomach Neoplasms; Gastrointestinal Neoplasms; Neoplasm Metastasis; Rectal Neoplasms | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Chemoembolization (Experimental): Chemoembolization with Irinotecan Bead in combination with Intravenous Chemotherapy Group (test arm)
  Interventions: Procedure: Chemoembolization with irinotecan Bead; Drug: Irinotecan
- Chemotherapy (Active Comparator): Irinotecan monotherapy: 250mg/m2 repeated every 3 weeks
  Interventions: Drug: Irinotecan

INTERVENTIONS:
Procedure: Chemoembolization with irinotecan Bead — Intra arterial chemoembolization using Irinotecan Bead 100mg irinotecan per procedure in combination with irinotecan monotherapy 250mg/m2 alternating on a 3 weekly schedule
  Other Names: Trans arterial Chemoembolization; Irinotecan Bead
  Arms: Chemoembolization
Drug: Irinotecan — Irinotecan monotherapy: 250mg/m2 repeated every 3 weeks
  Other Names: camptosar

SUMMARY:
The primary objective of this study is to evaluate the safety and efficacy of Irinotecan Bead in combination with intravenous chemotherapy versus intravenous chemotherapy alone in the treatment of unresectable liver metastases in patients with colorectal cancer. The results of this study are intended to be used in support of a PMA application for a combination device

DETAILED DESCRIPTION:
There are many treatments for metastatic colorectal cancer to the liver, and both the application and outcomes are highly dependant on the patients disposition. Whilst resection results in the best long term survival, it is often not a viable treatment option.

Irinotecan Bead is an embolization device intended to treat colorectal cancer metastases of the liver. As an adjunct to this, irinotecan is present in the microspheres which is released in a controlled manner into the local environment of the tumor. Irinotecan Bead is a combination of an approved embolization device and an approved chemotherapy agent. The device is a PVA based embolization agent from Biocompatibles UK Ltd, and the irinotecan is sourced from an FDA approved supplier.

Irinotecan, a topoisomerase inhibitor, was the first systemic chemotherapy drug other than 5-Fluorouracil (5-FU) to demonstrate significant activity in the treatment of metastatic colorectal cancer. Irinotecan is approved for use in combination with 5-FU/folinic acid in patients without prior chemotherapy, and for the second-line treatment of metastatic colorectal cancer as a single agent in patients who have failed an established 5-FU containing treatment regimen.

The purpose of this combination device as a treatment for cancer in the liver is twofold:

(i) Nutrient and oxygen starvation of the tumor. (ii) Minimization of chemotherapy wash-out with prolonged contact with tumor tissue.

Irinotecan Bead can be administered intra-arterially in the same manner as conventional TACE. The benefit of this product is that TACE is achieved in a simpler one-step procedure by precisely embolizing the arteries feeding the tumor, and as an ancillary action, the Irinotecan Bead may release a controlled dose of irinotecan into the tumor bed.

The potential benefits of Irinotecan Bead could be significant since a sustainable release of chemotherapy over time could have a greater effect on tumor mass, because optimal therapeutic efficacy of Irinotecan (an S phase-specific cytotoxic drug) generally requires prolonged exposure of the tumor to concentrations exceeding a minimum threshold.

Studies of low-dose, protracted administration of Irinotecan and other camptothecin analogues in mice bearing xenografts of human tumors have shown less toxicity and equal to or better antitumor activity than shorter, more intense dosing schedules. With the proposed device, the in-vivo and pre-clinical data shows that there is reduced systemic levels of Irinotecan, when delivered to tumorous tissue following embolization, and a longer, sustained concentration of the active metabolite, SN-38.

This is a multicentre, open labeled, prospective, randomized, controlled phase II study designed to assess the clinical performance of chemoembolization with Irinotecan Bead in combination with intravenous chemotherapy (irinotecan monotherapy) versus intravenous chemotherapy alone in the treatment of unresectable liver metastases in patients with colorectal cancer who previously failed first line chemotherapy.

The primary endpoint will be Progression Free Survival measured from the first treatment in this study until progression. Additional endpoints will be Pharmacokinetics of systemic Irinotecan and SN-38 (Irinotecan Bead treatment for feasibility group only); Tumor Response measured according to RECIST; Local tumor response (extent of necrosis in the treated lesions); hepatic progression free survival measured from first treatment until progression in the liver; change in tumor markers (CEA and optional CA19-9); performance status and overall survival assessed by telephone follow-up. Safety will be measured by assessing Adverse Events and Toxicity according to the NCI CTCAE v3.0 criteria.

Approximately 70 patients will be enrolled. The first 10 patients will be enrolled in a feasibility safety evaluation in the test arm of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of stage IV colorectal cancer with unresectable liver metastases (primary tumor may be present)
* Patients with at least one measurable liver metastases, with size > 1cm (RECIST criteria)
* Patients with liver dominant disease defined as ≥50% tumor body burden confined to the liver
* Patients with patent main portal vein
* Performance status ≤ 2 ECOG
* Life expectancy > 6 months
* Aged ≥18 years
* Patient has failed (discontinued for progression or toxicity) one prior line of chemotherapy for metastatic disease, preferably oxaliplatin-based (e.g. FOLFOX, CAPOX). Note that substitutions of oral versus IV 5-FU formulations, changes in 5-FU schedules, or discontinuations/re-starting of the same chemotherapy drugs will not be considered as separate lines of therapy, nor will the addition of "biologics" such as bevacizumab, cetuximab, or panitumumab
* Patient has no previous treatment with irinotecan
* At least 4 weeks since last administration of last chemotherapy and /or radiotherapy
* Hematologic function: ANC ≥ 1.5 x 109/L, platelets ≥75 x10-9/L, INR <1.5 (patients on therapeutic anticoagulants are not eligible)
* Adequate liver function as measured by: Total bilirubin ≤ 2.0mg/dl, ALT, AST ≤5 times ULN, albumin ≥2.5g/dl,
* Adequate renal function (creatinine ≤ 2.0mg/dl)
* Women of child bearing potential and fertile men are required to use effective contraception (negative serum βHCG/urine test for women of child-bearing age)
* Signed, written informed consent

Exclusion Criteria:

* Patient eligible for curative treatment (i.e. resection or radiofrequency ablation). Note: resectability is defined as a single tumor <5cm with adequate liver function defined: Total bilirubin ≤ 2.0mg/dl, ALT, AST ≤5 times ULN, albumin ≥2.5g/dl
* Contraindications to irinotecan:
* Chronic inflammatory bowel disease and/or bowel obstruction
* History of severe hypersensitivity reactions to irinotecan hydrochloride trihydrate, lactic acid or to any of the excipients of Camptosar
* Severe bone marrow failure
* History of Gilbert Syndrome (specific testing not required)
* Concomitant use with St John's Wort (Hypericum)
* Active bacterial, viral or fungal infection within 72 hours of study entry
* Women who are pregnant or breast feeding
* Previous irinotecan based therapy for metastatic disease
* Patients' whose only measurable disease is within an area of the liver previously subject to radiotherapy
* Allergy to contrast media that cannot be managed with standard care (e.g. steroids)
* Presence of another malignancy with the exception of cervical carcinoma in situ and stage I basal or squamous carcinoma of the skin
* Contraindicated for MRI or CT
* Patients previously treated with transarterial embolization (with or without chemotherapy)
* Any contraindication for hepatic embolization procedures:
* Large shunt as determined by the investigator (pretesting with TcMMA not required)
* Severe atheromatosis
* Hepatofugal blood flow
* Main portal vein occlusion (e.g. thrombus or tumor)
* Other significant medical or surgical condition, or any medication or treatment, that would place the patient at undue risk, that would preclude the safe use of chemoembolization or would interfere with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-12; Primary Completion 2011-01 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wells Messersmith, MD, Principal Investigator — University of Colorado, Denver
Locations (3):
- United States (3):
  - University of Colorado Cancer Center, Aurora, Colorado
  - Northwestern University, Chicago, Illinois
  - Lahey Clinic, Burlington, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chemoembolization | Chemotherapy
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemoembolization | Chemotherapy | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Full Range); unit: years] | 56 [55 to 57] | 63 [60 to 64] | 58.25 [55 to 64]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Time Frame: 1 year
Arm/Group | Chemoembolization | Chemotherapy
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Toxicity, Adverse Events and Serious Adverse Events (NCI CTCAE v3.0)
Description: 0 - No data collected
Time Frame: 6 weeks
Population: Data not collected study terminated early
Arm/Group | Chemoembolization | Chemotherapy
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Tumor Response (RECIST)
Time Frame: 1 year
Population: Study terminated ealry
Arm/Group | Chemoembolization | Chemotherapy
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Local Tumor Response (Extent of Necrosis in the Treated Lesions)
Time Frame: 1 year
Population: Study terminated ealry - data not collected
Arm/Group | Chemoembolization | Chemotherapy
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Hepatic Progression Free Survival
Description: Data not collected - study terminated ealry
Time Frame: 1 year
Population: Early termination - data not collected
Arm/Group | Chemoembolization | Chemotherapy
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Tumor Marker
Time Frame: 1 year
Population: Study terminated early. No Data collected
Arm/Group | Chemoembolization | Chemotherapy
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Performance Status (ECOG)
Description: No data collected
Time Frame: 1 year
Population: Study terminated early
Arm/Group | Chemoembolization | Chemotherapy
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Overall Survival
Time Frame: 1 year
Population: Study terminated ealry no data collected
Arm/Group | Chemoembolization | Chemotherapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 year
Description: No adverse events reported
Arm/Group | Chemoembolization | Chemotherapy
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days